CLINICAL TRIAL: NCT00507338
Title: A Phase 2 Study of an Aptameric Von Willebrand Factor Antagonist, ARC1779, in Patients With Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention
Brief Title: Study of ARC1779 in Patients With Acute Myocardial Infarction Undergoing PCI
Acronym: vITAL-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Archemix Corp. (Industry)
Responsible Party: James Gilbert, MD/Chief Medical Officer, Archemix, Corp.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARC1779-003
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Acute Myocardial Infarction
Keywords: percutaneous coronary intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ARC1779 low dose (Experimental): 0.1 mg/kg
  Interventions: Procedure: PCI
- ARC1779 mid dose (Experimental): 0.3 mg/kg
  Interventions: Procedure: PCI
- ARC1779 high dose (Experimental): 1.0 mg/kg
  Interventions: Procedure: PCI
- abciximab (Active Comparator): labeled regimen for primary PCI
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — early PCI for NSTEMI; primary PCI for STEMI

SUMMARY:
ARC1779 is a novel drug being tested in patients undergoing angioplasty and stenting as their primary treatment for heart attack.

DETAILED DESCRIPTION:
Adjunctive anti-thrombotic therapy for PCI of AMI may be improved by incorporation of a novel anti-platelet therapeutic principle, von Willebrand Factor antagonism. ARC1779 is a therapeutic oligonucleotide ("aptamer") which blocks the binding of the A1 domain of vWF to the platelet GPIb receptor, and thereby modulates platelet adhesion, activation, and aggregation under the high shear conditions of coronary arterial stenosis and plaque rupture. This study is intended to provide dose-ranging and clinical proof of concept for ARC1779 in a primary PCI population.

ELIGIBILITY:
Inclusion Criteria:

* troponin-positive NSTEMI, with diagnostic symptoms and/or ECG abnormalities present within the preceding 24 hours, and a planned "early invasive" management strategy
* STEMI, with planned primary PCI

Exclusion Criteria:

* History of bleeding diathesis or evidence of active abnormal bleeding within the previous 30 days
* Received treatment with fibrinolytic or GPIIb/IIIa antagonist drugs within the preceding 72 hours
* Received anticoagulant therapy with a low molecular weight heparin within the preceding 8 hours
* Severe hypertension (systolic blood pressure >200 mmHg or diastolic blood pressure >110 mmHg) not adequately controlled on antihypertensive therapy
* Major surgery or trauma within the preceding 6 weeks
* History of stroke within 30 days or any history of hemorrhagic stroke
* End-stage renal disease (ESRD) with dependency on renal dialysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
adequacy of reperfusion | 48 hours post-PCI

SECONDARY OUTCOMES:
bleeding | PCI to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gibson, MD, Study Chair — Harvard Medical School, Beth Israel Deaconess Medical Center; Franz-Josef Neumann, MD, Principal Investigator — Herz-Zentrum Bad Krozingen
Locations (1):
- Archemix Investigational Site, Saint Petersburg, Russia, Russia

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581